CLINICAL TRIAL: NCT03251638
Title: Neonatal Hearing Screening at Neonatal Intensive Care Unit of Assiut University Hospital
Brief Title: Neonatal Hearing Screening in Assiut Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nesma Gamal, Neonatal Hearing Screeing at Neonatal Intensive Care Unit of Assiut University Hospital, Assiut University
Other Study IDs: Assuit
Record Dates: First submitted 2017-08-12; First posted 2017-08-16 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Neonatal Hearing Impairment
Keywords: NHS( newborn hearing screening )

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hearing loss is one of the most common congenital anomalies. Early Intervention at or before 6 months of age allows a child with impaired hearing to develop normal speech and language.Auditory brainstem response , otoacoustic emissions testing have all been used in newborn hearing-screening programs

DETAILED DESCRIPTION:
Hearing loss is one of the most common congenital anomalies . It has been shown to be greater than that of most other diseases and syndromes (eg, phenylketonuria, sickle cell disease) screened at birth . Data from the newborn hearing-screening programs in Rhode Island, Colorado, and Texas showed that 2-4 of every 1000 neonates have hearing loss.

Early Intervention at or before 6 months of age allows a child with impaired hearing to develop normal speech and language, alongside his or her hearing peers and can prevent severe psychosocial, educational, and language impairment.( One of the most high risk population are neonates who spend time in the newborn intensive care unit, exposed to high frequency ventilation, hyperbilirubinemia, low birth-weight, and exposed to ototoxic medications.

Auditory brainstem response, otoacoustic emissions , and automated Auditory brainstem response testing have all been used in newborn hearing-screening programs. otoacoustic emissions are fast objective, efficient, and frequency-specific measurements of peripheral auditory sensitivity are used to assess response of the outer hair cells to acoustic stimuli. To measure otoacoustic emissions, a probe assembly is placed in the ear canal, tonal or click stimuli are delivered, and the otoacoustic emissions generated by the cochlea is measured with a microphone .

Currently, 2 types of evoked otoacoustic emissions measurements are used for newborn hearing screening: transient evoked otoacoustic emissions and distortion product otoacoustic emissions . Provided that the patient's middle ear function is normal, these measurements can be used to assess cochlear function for the 500-6000 Hz frequency range. The presence of evoked otoacoustic emissions responses indicates hearing sensitivity in the normal to near-normal range .

The Auditory brainstem response test records brainstem electrical activity in response to sounds presented to the infant via earphones. In contrast to the otoacoustic emissions test, the The Auditory brainstem response evaluates the auditory pathway from the external ear to the level of the brainstem, enabling diagnosis of auditory neuropathy, which is a less common cause of hearing impairment .

ELIGIBILITY:
Inclusion Criteria:

* A) Neonates of both sexes. (B) Neonates with the following risk factors according to the Joint Committee on Infant Hearing 2000 Position Statement:

  * In utero infection such as cytomegalovirus, rubella, toxoplasmosis, or herpes.
  * Neonatal indicators, specifically hyperbilirubinemia at a serum level requiring exchange transfusion, persistent pulmonary hypertension of the newborn associated with mechanical ventilation, and conditions requiring the use of extracorporeal membrane oxygenation
  * Low birth weight (1500-1800)grams

Exclusion Criteria:

* • Absence of high risk factors in the neonates.

Ages: 1 Day to 1 Month | Sex: All
Age Groups: Child
Study Population: Neonates who admitted at neonatal intensive care unit
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Neonatal hearing screening | 6months
  number of neonates who failed to pass emissions

CONTACTS AND LOCATIONS:
Overall Officials: Nafesa Hs Rafat, Prof, Study Director

REFERENCES:
- [Result] Connolly JL, Carron JD, Roark SD. Universal newborn hearing screening: are we achieving the Joint Committee on Infant Hearing (JCIH) objectives? Laryngoscope. 2005 Feb;115(2):232-6. doi: 10.1097/01.mlg.0000154724.00787.49. PMID 15689741
- [Result] Downs MP. Universal newborn hearing screening--the Colorado story. Int J Pediatr Otorhinolaryngol. 1995 Jul;32(3):257-9. doi: 10.1016/0165-5876(95)01183-c. PMID 7665273
- [Result] Erenberg A, Lemons J, Sia C, Trunkel D, Ziring P. Newborn and infant hearing loss: detection and intervention.American Academy of Pediatrics. Task Force on Newborn and Infant Hearing, 1998- 1999. Pediatrics. 1999 Feb;103(2):527-30. doi: 10.1542/peds.103.2.527. PMID 9925859
- [Result] Finitzo T, Albright K, O'Neal J. The newborn with hearing loss: detection in the nursery. Pediatrics. 1998 Dec;102(6):1452-60. doi: 10.1542/peds.102.6.1452. PMID 9832584
- [Result] Williams TR, Alam S, Gaffney M; Centers for Disease Control and Prevention (CDC). Progress in identifying infants with hearing loss-United States, 2006-2012. MMWR Morb Mortal Wkly Rep. 2015 Apr 10;64(13):351-6. PMID 25856256